CLINICAL TRIAL: NCT05891366
Title: Safety, Pharmacokinetics, and Pharmacodynamics of a Single, Ascending Dose of WAL0921 in Healthy Subjects
Brief Title: Single Ascending Dose Study of WAL0921 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Walden Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: WAL0921-01
Record Dates: First submitted 2023-05-20; First posted 2023-06-06 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WAL0921 (Experimental): Single intravenous infusion of investigational drug WAL0921
  Interventions: Drug: WAL0921
- Placebo (Placebo Comparator): Single intravenous infusion of normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WAL0921 — Investigational product WAL0921
  Arms: WAL0921
Drug: Placebo — Placebo product
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose study to evaluate the safety, pharmacokinetics, and pharmacodynamics of WAL0921 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, age ≥ 18 and ≤ 65 years at the time of anticipated dosing
2. Healthy individuals without known current or chronic medical conditions in the opinion of the Investigator
3. Body mass index (BMI) ≥ 18 and ≤ 32 kg/m2

Exclusion Criteria:

1. Clinically significant findings in physical examination, vital signs (blood pressure, heart rate, and body temperature), ECG, and safety laboratory parameters at screening in the opinion of the Investigator
2. Renal function calculated by the CKD-EPI (2021) equation with eGFR <90 mL/min/1.73 m2 at the time of screening
3. Abnormal levels of proteinuria detected on Urine Protein-Creatinine Ratio (UPCR) test >0.30 g/g
4. Any disease or condition that, in the opinion of the Investigator, might significantly compromise the cardiovascular, hematological, renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer) systems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Day 1 to Day 64

SECONDARY OUTCOMES:
Number of participants with clinically significant changes in hematology lab values | Day 64
  Hematology labs include complete blood count with differential and coagulation panel
Number of participants with clinically significant changes in chemistry lab values | Day 64
  Chemistry labs include a comprehensive metabolic panel
AUC | Day 1 to Day 64
  Area Under the Drug Concentration-Time Curve
Cmax | Day 1 to Day 64
  Maximum Observed Drug Concentration
Half-life | Day 1 to Day 64
  Drug terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Blair, MD, Study Director — Walden Biosciences, Inc.
Locations (1):
- PPD Pharmacology Unit, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No